CLINICAL TRIAL: NCT03154060
Title: Evaluation of the Accuracy and Precision of Flash Glucose Monitoring Sensors in Different Sites: the Abdomen and Upper Thigh Compared to the Upper Arm
Brief Title: Evaluation of the Accuracy and Precision of Flash Glucose Monitoring Sensors in Different Sites
Acronym: OUT OF SIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Onze Lieve Vrouwziekenhuis Aalst (Other)
Responsible Party: Principal Investigator, prof dr Pieter Gillard, Professor Doctor Pieter Gillard, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OOS-60146
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Flash glucose monitoring; Accuracy; Precision
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: open-label, prospective, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Using 3 Abbott FreeStyle Libre Flash Glucose Monitoring sensors in parallel and measure 7 times a day BG by capillary finger stick testing.
  Interventions: Device: Abbott FreeStyle Libre Flash Glucose Monitoring sensors

INTERVENTIONS:
Device: Abbott FreeStyle Libre Flash Glucose Monitoring sensors — Three FGM sensors will be inserted simultaneously (one on the back of the upper arm, abdomen and thigh) and will be worn for a consecutive 14 days. Throughout the study, patients should measure capillary blood glucose (BG) with the built-in BG meter of the Freestyle Libre at least 7 times per day (before and 1-2 hours after every meal and before bedtime). Additionally, patients should scan each sensor at least every 8 hours to obtain every measured interstitial glucose value. At the end visit (after 14 days), patients will come back to the hospital to download FGM and SMBG data.

SUMMARY:
On the first of July 2016, reimbursement for the Freestyle Libre Flash Glucose Monitoring (FGM) was introduced by the Belgian healthcare authority by means of a new diabetes convention. Making this the only way to receive the device in Belgium. Since then, many type 1 diabetes (T1D) patients switched to FGM. But some patients found the sensor on the upper arm too visible. Abbott does not recommend to place the sensor on a different place of the body than the back of the upper arm, because no tests were done yet (besides on the upper arm) to make an accuracy claim. With this study, we want to evaluate the accuracy and the precision of the Freestyle Libre FGM by using three FGM sensors simultaneously on different places of the body and perform regular self-monitoring of blood glucose (SMBG) tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of T1D for more than 6 months
* Adult patients ≥ 18 years
* Signed informed consent form

Exclusion Criteria:

* Pregnancy
* Patients with severe cognitive dysfunction or other disease which makes FGM use difficult.
* History of allergic reaction to any of the FGMs materials or adhesives when in contact with the skin.
* History of allergic reaction to chlorhexidine or alcohol anti-septic solution.
* Abnormal skin at the anticipated glucose sensor insertion sites (excessive hair, burn, inflammation, infection, rash, and/or tattoo).
* Presence of concomitant pathology that might cause edema at the insertion sites (such as heart failure, liver failure, kidney failure defined as eGFR < 45 ml/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Mean Absolute Relative Difference | 14 days
  Mean Absolute Relative Difference (MARD) between FGM measurements for the three insertion sites and paired SMBG measurements.

SECONDARY OUTCOMES:
Precision Absolute Relative Deviation | 14 days
  Precision Absolute Relative Deviation (PARD) between FGM measurements of the sensor on the back of the upper arm and paired FGM measurements of sensors on the abdomen and upper thigh.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Onze-Lieve-Vrouwziekenhuis Aalst, Aalst
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No